CLINICAL TRIAL: NCT00608283
Title: Live Kidney Donor Study (RELIVE-01)
Brief Title: Live Kidney Donor Study
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Health Resources and Services Administration (HRSA) (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: DAIT RELIVE-01
Record Dates: First submitted 2008-02-05; First posted 2008-02-06 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Kidney Transplantation; End Stage Renal Disease
Keywords: Kidney transplant; Live donor transplant
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Live Kidney Donors: People who are going to donate a kidney at one of the three transplant centers from August 2007 until June 2011

SUMMARY:
Kidney transplants from living donors now account for 40% of all the kidney transplants done in the United States. However, the current information on how donating a kidney can affect the donor's long term health needs further investigation. The purpose of this study is to collect data on a large number of live kidney donors and create and analyze a comprehensive database. Information about the number of living kidney donors, including those who have experienced kidney failure, heart problems, and death will be gathered for the database. Investigators will then use the database to identify the risks of kidney failure, associated conditions, and death after living donation. The database will also be used to identify characteristics that put donors at higher risk for health problems after donation.

DETAILED DESCRIPTION:
Kidney transplantation is the preferred treatment to dialysis for most people with kidney failure. However, the current waiting time to receive a kidney from a deceased donor is greater than 5 years in some parts of the United States. Kidneys from living donors have increased the number of kidneys available for transplantation and decreased the waiting period for those needing a transplant. Living kidney donation also provides several advantages over deceased donor kidneys, including more timely transplantation and longer function of the transplanted kidney. Despite these facts, there is inadequate information about whether living kidney donation may have serious adverse effects on the donor's health. Long-term data on the health risks of living donation are needed.

The purpose of this study is to establish and analyze a database of information on living donors who have or are going to donate a kidney at three transplant centers with longstanding live kidney donation programs through June 2011. Donor and recipient characteristics as well as specific data on kidney failure, heart disease, and death will be collected. National databases such as the Scientific Registry of Transplant Recipients, the Social Security Death Master File, the National Death Index and records maintained by the Centers for Medicare and Medicaid Services for patients with end stage renal disease (ESRD) will be used to supplement data provided by the participating transplant centers. After establishing the database, researchers expect to 1) determine the long-term risk of live kidney donation and 2) identify donor characteristics associated with higher risk for health problems after donation. Death, cause of death, and incidence of ESRD will be compared to those rates reported by the Centers for Disease Control and Prevention for the U.S. population during the same time period.

There will be no study visits for this study. Investigators will gather data from the medical charts of all live kidney donors from the three transplant centers through June 2011.

ELIGIBILITY:
Inclusion Criteria:

* Donated kidney at one of the three participating study centers

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People who will donate kidneys at one of the three transplant centers between August 2007 and June 2011
Sampling Method: Non-Probability Sample
Enrollment: 8951 (Actual)
Dates: Start 2007-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Overall mortality | Throughout study
Cause-specific mortality | Throughout study
End stage renal disease as defined in the protocol | Throughout study

SECONDARY OUTCOMES:
Cardiovascular and renal morbidity | Throughout study
6 months incidence of adverse events | At 6 months after kidney donation

CONTACTS AND LOCATIONS:
Overall Officials: Sandra J. Taler, MD, Principal Investigator — Division of Nephrology and Hypertension, Mayo Clinic; Clifton Kew, MD, Principal Investigator — University of Alabama at Birmingham; Hassan Ibrahim, MD, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Background] Baid-Agrawal S, Frei UA. Living donor renal transplantation: recent developments and perspectives. Nat Clin Pract Nephrol. 2007 Jan;3(1):31-41. doi: 10.1038/ncpneph0383. PMID 17183260
- [Background] Fehrman-Ekholm I, Norden G, Lennerling A, Rizell M, Mjornstedt L, Wramner L, Olausson M. Incidence of end-stage renal disease among live kidney donors. Transplantation. 2006 Dec 27;82(12):1646-8. doi: 10.1097/01.tp.0000250728.73268.e3. PMID 17198252
- [Background] Oien CM, Reisaeter AV, Leivestad T, Dekker FW, Line PD, Os I. Living donor kidney transplantation: the effects of donor age and gender on short- and long-term outcomes. Transplantation. 2007 Mar 15;83(5):600-6. doi: 10.1097/01.tp.0000255583.34329.dd. PMID 17353781
- [Result] Taler SJ, Messersmith EE, Leichtman AB, Gillespie BW, Kew CE, Stegall MD, Merion RM, Matas AJ, Ibrahim HN; RELIVE Study Group. Demographic, metabolic, and blood pressure characteristics of living kidney donors spanning five decades. Am J Transplant. 2013 Feb;13(2):390-8. doi: 10.1111/j.1600-6143.2012.04321.x. Epub 2012 Nov 8. PMID 23137211
- [Result] Jacobs CL, Gross CR, Messersmith EE, Hong BA, Gillespie BW, Hill-Callahan P, Taler SJ, Jowsey SG, Beebe TJ, Matas AJ, Odim J, Ibrahim HN; RELIVE Study Group. Emotional and Financial Experiences of Kidney Donors over the Past 50 Years: The RELIVE Study. Clin J Am Soc Nephrol. 2015 Dec 7;10(12):2221-31. doi: 10.2215/CJN.07120714. Epub 2015 Oct 13. PMID 26463883
- [Result] Jowsey SG, Jacobs C, Gross CR, Hong BA, Messersmith EE, Gillespie BW, Beebe TJ, Kew C, Matas A, Yusen RD, Hill-Callahan M, Odim J, Taler SJ; RELIVE Study Group. Emotional well-being of living kidney donors: findings from the RELIVE Study. Am J Transplant. 2014 Nov;14(11):2535-44. doi: 10.1111/ajt.12906. Epub 2014 Oct 7. PMID 25293374
- [Result] Gross CR, Messersmith EE, Hong BA, Jowsey SG, Jacobs C, Gillespie BW, Taler SJ, Matas AJ, Leichtman A, Merion RM, Ibrahim HN; RELIVE Study Group. Health-related quality of life in kidney donors from the last five decades: results from the RELIVE study. Am J Transplant. 2013 Nov;13(11):2924-34. doi: 10.1111/ajt.12434. Epub 2013 Sep 6. PMID 24011252
- [Result] Noppakun K, Cosio FG, Dean PG, Taler SJ, Wauters R, Grande JP. Living donor age and kidney transplant outcomes. Am J Transplant. 2011 Jun;11(6):1279-86. doi: 10.1111/j.1600-6143.2011.03552.x. Epub 2011 May 12. PMID 21564530
- [Result] Messersmith EE, Gross CR, Beil CA, Gillespie BW, Jacobs C, Taler SJ, Merion RM, Jowsey SG, Leichtman AB, Hong BA; RELIVE Study Group. Satisfaction With Life Among Living Kidney Donors: A RELIVE Study of Long-Term Donor Outcomes. Transplantation. 2014 Dec 27;98(12):1294-300. doi: 10.1097/TP.0000000000000360. PMID 25136843
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Heart, Lung, and Blood Institute (NHLBI) — https://www.nhlbi.nih.gov/
- Available data/document: Individual Participant Data Set: SDY289 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY289 — ImmPort study identifier is SDY289
- Available data/document: Study Protocol: SDY289 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY289 — ImmPort study identifier is SDY289
- Available data/document: Study summary, -design, -demographics, -files: SDY289 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY289 — ImmPort study identifier is SDY289